CLINICAL TRIAL: NCT00301275
Title: Assessing Free Immunoglobulin Light Chains in Patients With Myeloma
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: 2123
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2006-03-10 (Estimated); Status verified 2006-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Multiple myeloma is a disorder in which malignant plasma cells accumulate in the bone marrow. These plasma cells produce an abnormal protein called paraprotein / M spike in the serum which can be serially monitored to assess the response of tumour on therapy. The paraprotein has a heavy chain which can be either IgG, IgA, IgM or IgD and a light chain which can be either kappa or lambda.

At present, these can be assessed by serum and urine electrophoresis (SPE and UPE). These techniques are relatively insensitive and poorly quantitative compared with other immunoassays for tumour markers.

The potential of serum free light chain (flc) measurement as a marker for myeloma has been recognised for some time. However, development of such assays has proved elusive, primarily due to the difficulty in developing assays that are both convenient to use and have the required specificity to measure flc in serum. Recently , the assay has been standardised and is in use. Its likely that the assessment of flc might be a sensitive marker of documenting complete remission in patients with myeloma. The aim of this study is to study the flc in patients with myeloma in complete remission (CR) to see if patients have CR documented by standard criteria- are the free light chains still positive and if so are they better markers of remission. The samples will be collected and tested in batches of 60 each.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma patients in CR

Exclusion Criteria:

* not being able to give consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Ray Powles, FRCP, FRCpath, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS trust, Sutton, Surrey, United Kingdom